CLINICAL TRIAL: NCT02784249
Title: A Prospective, Randomized, Multi-Center, Open-Label Trial Comparing a Novel Goniotomy Procedure and an Ab Interno Trabecular Bypass Device in the Treatment of Mild to Moderate Glaucoma in Patients Undergoing Cataract Extraction
Brief Title: A Comparison of Two Ab Interno Procedures in the Treatment of Glaucoma in Patients Undergoing Cataract Extraction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New World Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C-16-04
Record Dates: First submitted 2016-05-24; First posted 2016-05-27 (Estimated); Last update posted 2021-07-14 (Actual); Status verified 2021-07

CONDITIONS: Open Angle Glaucoma
Keywords: Glaucoma; glaucoma surgery; ab interno
MeSH Terms: conditions — Glaucoma, Open-Angle; Glaucoma | interventions — Trabeculectomy; Cataract Extraction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Goniotomy (Experimental): Procedure: Goniotomy and trabecular excision in combination with planned cataract extraction via Phaco and PCIOL implant.
  Interventions: Procedure: Goniotomy; Procedure: Cataract Extraction
- Trabecular Micro-Bypass Stent (Active Comparator): Procedure: Device implantation in combination with planned cataract extraction via Phaco and PCIOL implant.
  Interventions: Device: Trabecular Micro-Bypass Stent; Procedure: Cataract Extraction

INTERVENTIONS:
Procedure: Goniotomy — Procedure: Goniotomy and trabecular excision with a novel ophthalmic knife in combination with planned cataract extraction via Phaco and PCIOL implant.
  Arms: Goniotomy
Device: Trabecular Micro-Bypass Stent — Procedure: Trabecular Micro-Bypass stent implantation in combination with planned cataract extraction via Phaco and PCIOL implant.
  Arms: Trabecular Micro-Bypass Stent
Procedure: Cataract Extraction — Cataract extraction via Phaco and PCIOL implant.

SUMMARY:
The purpose of this study is to compare the safety and efficacy of goniotomy performed with a novel ophthalmic knife compared to trabecular bypass stent implantation in mild to moderate glaucoma subjects who are also undergoing cataract extraction with phacoemulsification (Phaco) and posterior chamber intraocular lens (PCIOL) implant.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of open angle glaucoma (including pseudoexfoliation and pigmentary glaucoma)
* Diagnosis of mild to moderate glaucoma as defined by ICD-9 staging definitions 365.71 Mild/365.72 Moderate (including visual field defects and/or characteristic optic nerve abnormalities consistent with mild to moderate glaucoma)
* Planned removal of a visually significant cataract as determined by the Investigator (cortical, nuclear, subcapsular, or a combination) by manual phacoemulsification cataract extraction

Exclusion Criteria:

* Any glaucoma diagnosis other than those noted in inclusion criteria

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2016-06; Primary Completion 2017-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Percent reduction in mean IOP | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Luana Wilbur, BS, Study Director — Pilot to Pivotal Consulting, Inc.
Locations (1):
- Gundersen Health System, La Crosse, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No